CLINICAL TRIAL: NCT00530881
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Examine Safety and Establish Proof of Concept With PHX1149 in Patients With Type 2 Diabetes Mellitus
Brief Title: Randomized, Double-Blind, Placebo-Controlled, With PHX1149 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phenomix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX1149-Prot201
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 (Placebo Comparator)
  Interventions: Drug: PHX1149
- 3 active, 1 placebo (Placebo Comparator)
  Interventions: Drug: PHX1149

INTERVENTIONS:
Drug: PHX1149

SUMMARY:
This will be a 4-week, multicenter, randomized, double-blind, parallel group, placebo-controlled, safety, tolerability, and efficacy study. Patients will be screened and be on one of three doses of PHX1149 (a new drug candidate for the treatment of Type 2 diabetes ) or placebo. The drug is a "DPP4 inhibitor"

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treatment with metformin +/- TZD

Exclusion Criteria:

* Type 1 diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
postprandial blood glucose

SECONDARY OUTCOMES:
fasting blood glucose, HbA1c, safety

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Guler, MD, Study Director — Phenomix Corp.
Locations (1):
- Multiple Sites, San Diego, California, United States